CLINICAL TRIAL: NCT00757497
Title: Safety of Transcranial Direct Current Brain Stimulation (TDCS) for Improvement of Psychotic Symptoms and Cognitive Functioning in Childhood Onset Schizophrenia (COS)
Brief Title: Transcranial Direct Current Brain Stimulation to Treat Patients With Childhood-Onset Schizophrenia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 080211; 08-M-0211
Record Dates: First submitted 2008-09-20; First posted 2008-09-23 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2015-08-18

CONDITIONS: Childhood Onset Psychotic Disorders; Schizophrenia; Psychosis; Mental Disorders
Keywords: Treatment Study; Psychosis; Electrical Stimulation; Refractory; Novel; Childhood Onset Psychotic Disorders; Schizophrenia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mental Disorders

INTERVENTIONS:
Behavioral: Electrical Polarization

SUMMARY:
This study will test whether transcranial direct current stimulation (TDCS) can be used safely in children with schizophrenia and if it can improve memory and attention span or auditory hallucinations in these children, at least temporarily. TDCS has temporarily improved memory and attention span in healthy adults and a similar method called TMS has relieved auditory hallucinations in adults with schizophrenia. For the TDCS procedure, the child sits in a chair and two soft sponge electrodes are placed on the child s forehead and held in place with a soft wrapping. One sponge electrode is placed on an arm. The electrodes are attached to a stimulator with a wire.

Children with schizophrenia who meet the following criteria may be eligible for this study:

* Are 10 yrs or older age.
* Are participating in NIH protocol 03-M-0035.
* Are on a stable medication regimen for at least 6 months.
* Have problems with memory and attention span or have auditory hallucinations.

Participants are randomly assigned to receive either real or sham TDCS on an inpatient or outpatient basis in 20-minute sessions daily, except weekends, for 10 days. For real TDCS, patients receive stimulation to the front of the brain. For sham stimulation, the children have electrodes placed on the forehead, but no actual stimulation is delivered. In addition to TDCS, patients have the following procedures:

* Checks of blood pressure, pulse and breathing rate before, during and right after each stimulation and again 8 hours later.
* Electrocardiogram (EKG) and electroencephalogram (EEG) before starting stimulation and after completing the 10 days of TDCS.
* Interviews and examinations to check for side effects of TDCS.
* Pen-and-paper or computer tests of learning, attention and memory.
* At the end of the 10 sessions, children who were in the sham TDCS group are offered the same number of sessions of active TDCS.
* Follow-up telephone call 1 month after the end of stimulation to see how the child is doing.
* 1- to 2-day outpatient visit 6 months after the stimulation. This visit includes interviews with the parent and the child, rating of the child s psychiatric symptoms, and pen-and-paper or computer tests of thinking, attention and memory.

DETAILED DESCRIPTION:
Background: The majority (about 75%) of patients with childhood onset schizophrenia still have impairing cognitive and psychotic symptoms after drug treatment optimization. Recent studies with transcranial magnetic stimulation (TMS) indicate moderate efficacy in symptom reduction in adult patients with schizophrenia. Transcranial direct current stimulation (TDCS) may be a safe and effective additional treatment of residual symptoms of schizophrenia in medication stable patients. Recent research into adult-onset schizophrenia established both safety and efficacy in 20-minute daily DC polarization (TDSC).

Objective: To establish whether bilateral DC polarization (using TDCS) of either dorsolateral prefrontal cortex or superior temporal cortex is safe in patients with childhood onset schizophrenia and whether it is associated with improvement in cognitive performance or reduction in auditory hallucination (psychotic symptoms) respectively.

Study population: Up to 40 patients with schizophrenia, ages 10 and older will be recruited. All patients will be on optimized medications for at least 2 months prior to this study.

Design: The design has two concurrent study options; both double-blind sham controlled, with 10-day, 40-minute daily DC polarization. Patients will be selected for one of the two treatment options: 1. Bilateral Anodal DC polarization of prefrontal cortex or 2. Bilateral Cathodal DC polarization of superior temporal cortex. A small battery powered device (Phoresor II Auto Model PM850) approved by the FDA for iontophoretic transdermal drug delivery will be used to administer the DC current. Sham treatment will be electrode placement without current.

Outcome Measures: The primary outcome measure would be to determine whether TDCS treatment is safe in children and adults with schizophrenia, as assessed by vital signs monitoring, reporting/evaluation of adverse effects, clinical ratings and neurocognitive performance.

Secondary outcome measures: The secondary outcome measures would be improvement on 1) Hallucination Change Scale (HCS) and Auditory Hallucinations Rating Scale (AHRS) for auditory hallucinations; SAPS, SANS and BPRS scales for psychotic symptoms and 2) performance on the working memory (verbal and non verbal), attention/vigilance, and verbal learning sub tests for cognitive improvement.

Exploratory Measure: Effect of DC polarization on regional GM cortical thickness in DLPFC and STG regions.

ELIGIBILITY:
* INCLUSION CRITERIA:

COS patients (age 10 and above) recruited and followed under the current protocol 03-M-0035, where subjects have been stable (in the judgment of the investigator) on their medications for 2 months with or without PRN medications but continue to experience either:

1. Cognitive difficulties as evidenced by information from parents and teachers, clinical interview, and performance (below average based on published norms for each test) on neurocognitive tests (WMS-III Spatial Span (nonverbal) and WMS-III Letter-Number Sequencing (verbal) attention/vigilance (CPT-IP), and verbal learning (HVLT-R), all sub tests of the NIMH MATRICS battery).
2. Significant auditory hallucinations as measured by SAPS (scores above 2) or BPRS (scores above 3).

EXCLUSION CRITERIA:

In addition to the exclusion criteria under protocol 03-M-0035, the following will be exclusionary:

1. Broken or abnormal skin in the area of the electrodes.
2. Presence of metal in the cranial cavity.
3. Holes in the skull from trauma or surgery.
4. Positive pregnancy test.
5. Presence of other psychiatric illness (e.g. severe anxiety, OCD etc) unless the patient has been on stable medication for the prior 2 months

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09-17; Study Completion 2015-08-18 (Actual)

PRIMARY OUTCOMES:
TDCS treatment is safe in childhood onset schizophrenia

SECONDARY OUTCOMES:
Improvement in cognition and psychosis

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Gogtay, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Asarnow JR, Ben-Meir S. Children with schizophrenia spectrum and depressive disorders: a comparative study of premorbid adjustment, onset pattern and severity of impairment. J Child Psychol Psychiatry. 1988 Jul;29(4):477-88. doi: 10.1111/j.1469-7610.1988.tb00738.x. PMID 3215919
- [Background] Watkins JM, Asarnow RF, Tanguay PE. Symptom development in childhood onset schizophrenia. J Child Psychol Psychiatry. 1988 Nov;29(6):865-78. doi: 10.1111/j.1469-7610.1988.tb00759.x. PMID 3235494
- [Background] Russell AT, Bott L, Sammons C. The phenomenology of schizophrenia occurring in childhood. J Am Acad Child Adolesc Psychiatry. 1989 May;28(3):399-407. doi: 10.1097/00004583-198905000-00017. PMID 2738007
- [Derived] Berman RA, Gotts SJ, McAdams HM, Greenstein D, Lalonde F, Clasen L, Watsky RE, Shora L, Ordonez AE, Raznahan A, Martin A, Gogtay N, Rapoport J. Disrupted sensorimotor and social-cognitive networks underlie symptoms in childhood-onset schizophrenia. Brain. 2016 Jan;139(Pt 1):276-91. doi: 10.1093/brain/awv306. Epub 2015 Oct 22. PMID 26493637